CLINICAL TRIAL: NCT03235414
Title: Determination of Normal Liver Stiffness by MR Elastography in Children
Brief Title: Normal Liver Stiffness by MR Elastography
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Massachusetts General Hospital (Other); Washington University School of Medicine (Other); Children's Hospital of Philadelphia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CIN001-Liver stiffness
Record Dates: First submitted 2017-07-28; First posted 2017-08-01 (Actual); Results first posted 2020-08-27 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-07

CONDITIONS: Liver Diseases
MeSH Terms: conditions — Liver Diseases | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Normals (Experimental): Will receive an MRI and a blood draw
  Interventions: Device: MRI; Diagnostic Test: Blood draw

INTERVENTIONS:
Device: MRI — Will receive a one time research MRI (MR elastography)
Diagnostic Test: Blood draw — Will receive a one time blood draw to confirm healthy liver status

SUMMARY:
Healthy children will be recruited to under Magnetic Resonance Imaging (MRI)along with MR elastography to determine normal liver stiffness values.

DETAILED DESCRIPTION:
MR elastography (MRE) is playing a growing role in the non-invasive diagnosis and monitoring of liver disease in the pediatric population. There is, however, little data specific to the use of this technique in children with existing data and techniques largely extrapolated from adult studies. Existing studies suggest that liver stiffness values may be different between children and adults [Etchell, Xanthakos]. As such there is an unmet need for uniquely pediatric data in both healthy and diseased cohorts. To address the need for such data, the investigators plan a multi-site, prospective study of healthy pediatric (<18 years of age) volunteers to determine normal liver stiffness measured by MR elastography across the range of MRI equipment.

ELIGIBILITY:
Inclusion Criteria:

* Age 7-17 years
* No documented history of liver diseases
* English speaking

Exclusion Criteria:

* NPO less than 4 hours
* Body mass index <10th or > 85th percentile for age
* Documented history of liver disease
* Pregnancy
* Inability to lie still for duration of the MRI
* Inability to breath hold for the duration of the 15-20 second MR elastography sequence
* Standard contraindication to MRI (implanted hardware, etc.)
* Requirement of sedation or general anesthesia for MRI
* Abnormality of any measured liver function test
* Liver fat fraction >5% by MRI PDFF

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 101 (Actual)
Dates: Start 2018-02-19 (Actual); Primary Completion 2020-06-25 (Actual); Study Completion 2020-07-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Trout, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Trout AT, Anupindi SA, Gee MS, Khanna G, Xanthakos SA, Serai SD, Baikpour M, Calle-Toro JS, Ozturk A, Zhang B, Dillman JR. Normal Liver Stiffness Measured with MR Elastography in Children. Radiology. 2020 Dec;297(3):663-669. doi: 10.1148/radiol.2020201513. Epub 2020 Sep 22. PMID 32960728

RESULTS

PARTICIPANT FLOW:
Groups:
- Normals: Healthy participants receive an MRI and a blood draw
  MRI: Will receive a one time research MRI (MR elastography)
  Blood draw: Will receive a one time blood draw to confirm healthy liver status
Period: Overall Study
Arm/Group | Normals
Started | 101
Completed | 101
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Healthy Participants-Of the 101 participants enrolled 78 had no exclusionary data after completion of the single time point study. 7 had missing data
Arm/Group | Normals
Number analyzed (Participants) | 71
Age, Categorical [Count of Participants; unit: Participants] — Population: Healthy Participants-Of the 101 participants enrolled 78 had no exclusionary data after completion of the single time point study. 7 had missing data
  Participants
    <=18 years | 71
    Between 18 and 65 years | 0
    >=65 years | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] — Population: Healthy Participants-Of the 101 participants enrolled 78 had no exclusionary data after completion of the single time point study. 7 had missing data
  years | 12 [10 to 15]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Healthy Participants-Of the 101 participants enrolled 78 had no exclusionary data after completion of the single time point study. 7 had missing data
  Participants
    Female | 39
    Male | 32
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 71

OUTCOME MEASURES:

1. Primary Outcome: Liver Stiffness
Description: Liver stiffness is a measure of a mechanical property of tissue (stiffness). This can be measured non-invasively by MR elastography, a technique that involves applying an external vibration to the abdomen and measuring the progression of shear waves through the underlying liver using MRI.
  Purpose of the study was to determine normal (healthy) liver stiffness as measured by MRE
Time Frame: During investigation
Population: as for baseline characteristics
Measure: Median (Inter-Quartile Range); unit: kPa
Groups:
- Healthy Participants: Healthy participants will undergo Magnetic Resonance Elastography Imaging of the liver
Arm/Group | Healthy Participants
Number analyzed (Participants) | 71
kPa | 2.1 [1.9 to 2.3]

2. Secondary Outcome: Cross-platform Variability
Description: To assess for cross-platform (different MRI vendors) variability in normal MRI liver stiffness values
Time Frame: During Investigation
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: kPa
Arm/Group | Healthy Participants
Number analyzed (Participants) | 71
kPa
  GE | 2.1 (0.5)
  Philips | 2.3 (0.4)
  Siemens | 2.1 (0.2)

3. Secondary Outcome: Cross-field Strength
Description: To assess cross-field strength (1.5T vs. 3T) variability in normal MRI liver stiffness values
Time Frame: During investigation
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: kPa
Arm/Group | Healthy Participants
Number analyzed (Participants) | 71
kPa
  1.5T | 2.3 (0.4)
  3T | 2.1 (0.4)

4. Secondary Outcome: Sex-related Differences
Description: To assess for sex-related (male vs. female) differences in normal MRI liver stiffness values
Time Frame: During investigation
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: kPa
Arm/Group | Healthy Participants
Number analyzed (Participants) | 71
kPa
  Female | 2.2 (0.4)
  Male | 2.2 (0.4)

ADVERSE EVENTS:
Time Frame: During investigation
Arm/Group | Healthy Participants
All-Cause Mortality (participants affected / at risk) | 0/101
Serious Adverse Events (participants affected / at risk) | 0/101
Other Adverse Events (participants affected / at risk) | 0/101

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-04-18): https://cdn.clinicaltrials.gov/large-docs/14/NCT03235414/Prot_SAP_000.pdf
  • Informed Consent Form (2018-07-30): https://cdn.clinicaltrials.gov/large-docs/14/NCT03235414/ICF_001.pdf